CLINICAL TRIAL: NCT04472936
Title: Long-term outcomeS of cavotrIcuspid isthMus-dePendent fLuttEr Ablation: Randomized Study Comparing Single vs Double Catheter Procedure
Brief Title: Long-term outcomeS of cavotrIcuspid isthMus-dePendent fLuttEr Ablation: Single vs Double Catheter Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Research Coordinator of the Heart Institute, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIMPLE
Record Dates: First submitted 2020-06-13; First posted 2020-07-16 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Atrial Flutter
Keywords: Atrial flutter; Catheter ablation; Single catheter approach
MeSH Terms: conditions — Atrial Flutter

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Double venous femoral access will be obtained. A duodecapolar catheter placed around tricuspid annulus will be used to prove isthmus block after CTI ablation.
  Interventions: Procedure: Traditional approach
- Group B (Experimental): Ablation will be performed similar as described in the Group A. After the ablation line is over, PRI on the surface ECG will be used to prove isthmus block after CTI ablation.
  Interventions: Procedure: Single catheter approach

INTERVENTIONS:
Procedure: Single catheter approach — Single venous femoral access will be obtained and the ablation will be performed similar to Group A. After the ablation line is over, we will confirm CTI block using the PRI. During atrial pacing (10 V, 1.5 ms) at a stable cycle length (range 500-700ms) from the tip of the ablation catheter with a sweep speed of 300mm/s, the ablation catheter will be placed first at 5 o'clock (medial to CTI line), then at 7 o'clock (lateral to CTI line), and finally at 9 o'clock position, and the corresponding PRIs will be measured for each pacing site. CTI block is assumed when: (i) the PRI at 7 o'clock is >80ms longer than that at pacing sites of 5, and (ii) the PRI at 9 o'clock is shorter than the PRI at 7 o'clock.
  Arms: Group B
Procedure: Traditional approach — Double venous femoral access will be obtained. A duodecapolar catheter will be positioned in the right atrium around the tricuspid valve annulus (TVA) to record activation sequence around the tricuspid annulus. An ablation catheter will be positioned using fluoroscopic guidance in the central CTI, 6 o'clock in a left anterior oblique view. The distal ablation electrode position will then be adjusted toward or away from the TVA, based on the ratio of atrial and ventricular electrogram amplitudes with an optimal ratio of 1:2 or 1:4 at the TVA. After the ablation catheter is positioned, it will be very slowly withdrawn during ablation toward the inferior vena cava while radiofrequency energy is applied continuously. CTI block will be evaluated after ablation by determining the right atrial activation sequence during pacing from the low lateral right atrium and coronary sinus ostium.
  Arms: Group A

SUMMARY:
Catheter ablation is recommended as first-line therapy for most patients with typical atrial flutter. The most common approach is to create an ablation line across the cavotricuspid isthmus (CTI). Traditionally, atrial flutter ablation has been performed with a conventional approach using two catheters, an ablation catheter and a duodecapolar catheter that is placed at the level of the tricuspid annulus to confirm the CTI block. Recently, a single catheter approach has been described using the behavior of PR interval change during differential pacing over the ablation line to prove CTI block. This prospective, randomized, multicenter study analyzes the effectivity of a single catheter approach compared with conventional approach in terms of clinical outcomes.

DETAILED DESCRIPTION:
Typical atrial flutter is a reentrant rhythm in the right atrium that is constrained anteriorly by the tricuspid annulus and posteriorly by the crista terminalis and eustachian ridge. Catheter ablation is the first-line therapy for most patients with typical atrial flutter. The most common approach is to create an ablation line across the CTI, from the tricuspid annulus to the inferior vena cava. Traditionally, atrial flutter ablation has been performed with a conventional approach using two catheters, an ablation catheter and a duodecapolar catheter that is placed at the level of the tricuspid annulus that allows to evaluate the right atrial activation sequence to confirm the CTI block. Recently, a single catheter approach has been described using the behavior of PR interval (PRI) change during differential pacing over the ablation line to prove CTI block. The PRIs is measured for three different pacing site, 5 o'clock (medial to CTI line), 7 o'clock (lateral to CTI line), and 9 o'clock position. CTI block was assumed when the PRI at 7 o'clock was >80ms longer than that at pacing sites of 5 o'clock and the PRI at 9 o'clock was shorter than the PRI at 7 o'clock. However, a direct comparison between this approach and the conventional one was not yet performed. This prospective, randomized, multicenter study analyzes the effectivity of a single catheter approach compared with conventional approach in terms of clinical outcomes. Our research hypothesis is that a single catheter approach has the possible advantages of being a faster, more efficient and cheaper procedure than the conventional approach. Moreover, as it only requires a single venous access, the risk of complications is decreased.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at any of the centers to perform a CTI ablation.
* Signed informed consent

Exclusion Criteria:

* Age < 18 years.
* Pregnancy.
* Impossibility to perform CTI ablation.
* Impossibility to measure PRI (complete atrioventricular block).
* Ablation of other cardiac arrhythmias during the same procedure.
* Medical, geographical and social factors that make study participation impractical, and inability to give written informed consent. Patient's refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2020-07-16 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Clinical outcomes | 6 months
  The recurrence rate of typical atrial flutter at 6 months post cavotricuspid isthmus ablation will be evaluated in both groups to determine if the single catheter approach is non-inferior when compared to traditional approach using two catheters.

SECONDARY OUTCOMES:
Efficiency in total procedure time | 6 months
  The total procedure time time will be measured in both groups to determine if the single catheter approach is more efficient procedure.
Efficiency in ablation time | 6 months
  The ablation time will be measured in both groups to determine if the single catheter approach is more efficient procedure.
Efficiency in fluoroscopy time | 6 months
  The fluoroscopy time will be measured in both groups to determine if the single catheter approach is more efficient procedure.
Complications | 6 months
  We will compare the complication rate of both approaches.
Cost-effectiveness | 6 months
  We will perform a cost-effectiveness analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Berruezo, MD, PhD, Principal Investigator — Centro Medico Teknon
Locations (3):
- Spain (3):
  - Centro Medico Teknon, Barcelona
  - Puerta del Mar University Hospital, Cadiz
  - Virgen del Rocio University Hospital, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Feld GK, Fleck RP, Chen PS, Boyce K, Bahnson TD, Stein JB, Calisi CM, Ibarra M. Radiofrequency catheter ablation for the treatment of human type 1 atrial flutter. Identification of a critical zone in the reentrant circuit by endocardial mapping techniques. Circulation. 1992 Oct;86(4):1233-40. doi: 10.1161/01.cir.86.4.1233. PMID 1394929
- [Background] Cosio FG, Lopez-Gil M, Goicolea A, Arribas F, Barroso JL. Radiofrequency ablation of the inferior vena cava-tricuspid valve isthmus in common atrial flutter. Am J Cardiol. 1993 Mar 15;71(8):705-9. doi: 10.1016/0002-9149(93)91014-9. PMID 8447269
- [Background] Lesh MD, Van Hare GF, Epstein LM, Fitzpatrick AP, Scheinman MM, Lee RJ, Kwasman MA, Grogin HR, Griffin JC. Radiofrequency catheter ablation of atrial arrhythmias. Results and mechanisms. Circulation. 1994 Mar;89(3):1074-89. doi: 10.1161/01.cir.89.3.1074. PMID 8124793
- [Background] Page RL, Joglar JA, Caldwell MA, Calkins H, Conti JB, Deal BJ, Estes NA III, Field ME, Goldberger ZD, Hammill SC, Indik JH, Lindsay BD, Olshansky B, Russo AM, Shen WK, Tracy CM, Al-Khatib SM. 2015 ACC/AHA/HRS guideline for the management of adult patients with supraventricular tachycardia: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Heart Rhythm. 2016 Apr;13(4):e136-221. doi: 10.1016/j.hrthm.2015.09.019. Epub 2015 Sep 25. No abstract available. PMID 26409100
- [Background] Shah DC, Takahashi A, Jais P, Hocini M, Clementy J, Haissaguerre M. Local electrogram-based criteria of cavotricuspid isthmus block. J Cardiovasc Electrophysiol. 1999 May;10(5):662-9. doi: 10.1111/j.1540-8167.1999.tb00243.x. PMID 10355922
- [Background] Madaffari A, Krisai P, Spies F, Knecht S, Schaer B, Kojic D, Kuhne M, Sticherling C, Osswald S. Ablation of typical atrial flutter guided by the paced PR interval on the surface electrocardiogram: a proof of concept study. Europace. 2019 Nov 1;21(11):1750-1754. doi: 10.1093/europace/euz208. PMID 31384937
- [Background] Calkins H, Canby R, Weiss R, Taylor G, Wells P, Chinitz L, Milstein S, Compton S, Oleson K, Sherfesee L, Onufer J; 100W Atakr II Investigator Group. Results of catheter ablation of typical atrial flutter. Am J Cardiol. 2004 Aug 15;94(4):437-42. doi: 10.1016/j.amjcard.2004.04.058. PMID 15325925